CLINICAL TRIAL: NCT03996343
Title: Laryngeal Mask Airway Versus Endotracheal Intubation for Airway Management During General Anesthesia in Obese Children
Brief Title: Airway Management and Weight in Children
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Investigator leaving institution
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Olubukola Nafiu, Associate Professor of Anesthesiology, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: HUM00132290
Record Dates: First submitted 2019-06-20; First posted 2019-06-24 (Actual); Last update posted 2019-06-24 (Actual); Status verified 2019-06

CONDITIONS: Perioperative Respiratory Adverse Events; Airway Management
Keywords: Laryngeal mask airway; Endotracheal intubation; Obese
MeSH Terms: conditions — Obesity | interventions — Intubation, Intratracheal; Laryngeal Masks

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Endotracheal intubation (Experimental)
  Interventions: Device: Endotracheal intubation
- Laryngeal mask airway (Experimental)
  Interventions: Device: Laryngeal mask airway

INTERVENTIONS:
Device: Endotracheal intubation — COMPLETE
  Arms: Endotracheal intubation
Device: Laryngeal mask airway — COMPLETE
  Arms: Laryngeal mask airway

SUMMARY:
The investigators in this study want to see how overweight/obese children who undergo elective surgery requiring airway management react to general anesthesia. They believe that the incidence of perioperative respiratory adverse events (PRAE) associated with Laryngeal mask airway (LMA) use during general anesthesia in overweight/obese children is lower than that associated with endotracheal intubation (ETT).

ELIGIBILITY:
Inclusion Criteria:

* sex-specific body mass index (BMI) is ≥85th percentile
* elective surgical outpatient peripheral or lower abdominal procedures
* Surgery length estimated to last between 30 and 120 minutes

Exclusion Criteria:

* Active gastro-esophageal reflux, possible difficult intubation or planned asleep fiber optic intubation, cardiac disease, thoracic deformities, upper abdominal, and thoracic or airway surgeries.
* Children with active asthmatic attack or those considered to be "full stomach" will also be excluded.
* Laparoscopic surgical procedures and those requiring extreme head-down tilt will also be excluded.
* Children with a physiology or other condition requiring a certain type of airway for the procedure will also be excluded
* Children whose anesthesiologist is not agreeable to randomization of airway management choice will also be excluded.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2019-05 (Estimated); Primary Completion 2021-06 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Severe respiratory adverse events | perioperative period
  laryngospasm, bronchospasm

CONTACTS AND LOCATIONS:
Overall Officials: Olubukola Nafiu, MD, Principal Investigator — University of Michigan
Locations (1):
- The University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No